CLINICAL TRIAL: NCT00233285
Title: Factors in Childhood Lung Susceptibility to Pollution
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1306; R01HL061768 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2009-04

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

SUMMARY:
To investigate gene-environment interactions that may influence susceptibility to respiratory illness in children living in highly polluted areas in California.

DETAILED DESCRIPTION:
BACKGROUND:

Ambient air pollutants and tobacco smoke produce adverse respiratory health effects in children. Differences in susceptibility for these outcomes are likely to involve genetic variation in multiple pathophysiological pathways that modulate responses and subsequent biologic effects following exposure. The study initially investigated the hypothesis that genetic variants in oxidant stress pathways modulate the occurrence of adverse outcomes using a candidate gene approach in the Children's Health Study (CHS), a longitudinal study of children's respiratory health in 12 Southern California communities. The investigators found that variants in GSTM1 (null), GSTP1 (A105G), TNF (- 308), and ICAM-1 (241) were associated with reduced lung function growth, increased asthma occurrence, and increased respiratory illnesses. These variants also showed gene-environment and gene-gene interactions with tobacco smoke and ambient air pollutants. Their findings add to the growing body of evidence that pathways involving glutathione (GSH) play important roles in respiratory health.

DESIGN NARRATIVE:

In the initial grant period, the investigators studied the effects of ambient air pollution and tobacco smoke on children's respiratory health and the role of diet, physical activity and genetic variation on susceptibility to ambient air pollutants and completed each of the specific aims. They noted associations between genotypes studied and reduced lung function growth, increased sensitivity to in utero exposure to maternal smoking, increased the risk of asthma, and risk of respiratory-related school absences, varied by GSTM1 and GSTP1 genotype. They noted that diets low in antioxidant vitamins were associated with deficits in lung function and that low magnesium intake was associated with lung function deficits. Finally, the investigators identified haplotype structure and tag single nucleotide polymorphisms (SNPs) for selected candidate loci and employed a limited version of haplotype analysis for investigation of association of three ICAM-1 variants on childhood asthma.

The investigators will extend their candidate gene association study using existing data from the Children's Health Study (CHS), to examine the role of sequence variation in 38 genes in five glutathione (GSH) pathways including GSH production, transport, and redox cycling, electrophil and oxidation products detoxification, and nitric oxide cell signaling. The exposures of interest are ozone (O3), nitric oxide (NO2), ambient PM2.5, and tobacco smoke. The respiratory health outcomes are lung function growth, asthma, and respiratory absences. Associations of respiratory health outcomes with sequence variants in candidate genes and air pollution will be assessed using haplotypes and functional SNPs. They will test for overall association of a locus with outcomes using functional SNPs and a haplotype-based approach, and gene-gene and gene-environment interaction within and between pathways will also be examined using approaches to minimize multiple comparisons issues. Confounding by admixture will be addressed using SNP-based genome-wide control methods. Finally, hierarchical Bayesian models of these complex pathways incorporate a priori knowledge about biological relationships to efficiently examine interactions within and between pathways.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gilliland — University of Southern California

REFERENCES:
- [Background] Gilliland FD, Li YF, Saxon A, Diaz-Sanchez D. Effect of glutathione-S-transferase M1 and P1 genotypes on xenobiotic enhancement of allergic responses: randomised, placebo-controlled crossover study. Lancet. 2004 Jan 10;363(9403):119-25. doi: 10.1016/S0140-6736(03)15262-2. PMID 14726165
- [Background] Wenten M, Berhane K, Rappaport EB, Avol E, Tsai WW, Gauderman WJ, McConnell R, Dubeau L, Gilliland FD. TNF-308 modifies the effect of second-hand smoke on respiratory illness-related school absences. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1563-8. doi: 10.1164/rccm.200503-490OC. Epub 2005 Sep 15. PMID 16166621
- [Background] Li YF, Tsao YH, Gauderman WJ, Conti DV, Avol E, Dubeau L, Gilliland FD. Intercellular adhesion molecule-1 and childhood asthma. Hum Genet. 2005 Sep;117(5):476-84. doi: 10.1007/s00439-005-1319-7. Epub 2005 Jul 14. PMID 16021473
- [Background] Li YF, Langholz B, Salam MT, Gilliland FD. Maternal and grandmaternal smoking patterns are associated with early childhood asthma. Chest. 2005 Apr;127(4):1232-41. doi: 10.1378/chest.127.4.1232. PMID 15821200
- [Background] Salam MT, Li YF, Langholz B, Gilliland FD; Children's Health Study. Early-life environmental risk factors for asthma: findings from the Children's Health Study. Environ Health Perspect. 2004 May;112(6):760-5. doi: 10.1289/ehp.6662. PMID 15121522
- [Background] Gilliland FD, Berhane KT, Li YF, Gauderman WJ, McConnell R, Peters J. Children's lung function and antioxidant vitamin, fruit, juice, and vegetable intake. Am J Epidemiol. 2003 Sep 15;158(6):576-84. doi: 10.1093/aje/kwg181. PMID 12965883
- [Background] Gilliland FD, Berhane K, Islam T, McConnell R, Gauderman WJ, Gilliland SS, Avol E, Peters JM. Obesity and the risk of newly diagnosed asthma in school-age children. Am J Epidemiol. 2003 Sep 1;158(5):406-15. doi: 10.1093/aje/kwg175. PMID 12936895
- [Background] Gilliland FD, Berhane K, Islam T, Wenten M, Rappaport E, Avol E, Gauderman WJ, McConnell R, Peters JM. Environmental tobacco smoke and absenteeism related to respiratory illness in schoolchildren. Am J Epidemiol. 2003 May 15;157(10):861-9. doi: 10.1093/aje/kwg037. PMID 12746237
- [Background] Gilliland FD, Berhane K, Li YF, Rappaport EB, Peters JM. Effects of early onset asthma and in utero exposure to maternal smoking on childhood lung function. Am J Respir Crit Care Med. 2003 Mar 15;167(6):917-24. doi: 10.1164/rccm.200206-616OC. Epub 2002 Dec 12. PMID 12480608
- [Background] Xie B, Gilliland FD, Li YF, Rockett HR. Effects of ethnicity, family income, and education on dietary intake among adolescents. Prev Med. 2003 Jan;36(1):30-40. doi: 10.1006/pmed.2002.1131. PMID 12473422
- [Background] Gilliland FD, Li YF, Dubeau L, Berhane K, Avol E, McConnell R, Gauderman WJ, Peters JM. Effects of glutathione S-transferase M1, maternal smoking during pregnancy, and environmental tobacco smoke on asthma and wheezing in children. Am J Respir Crit Care Med. 2002 Aug 15;166(4):457-63. doi: 10.1164/rccm.2112064. PMID 12186820
- [Background] Gilliland FD, Rappaport EB, Berhane K, Islam T, Dubeau L, Gauderman WJ, McConnell R. Effects of glutathione S-transferase P1, M1, and T1 on acute respiratory illness in school children. Am J Respir Crit Care Med. 2002 Aug 1;166(3):346-51. doi: 10.1164/rccm.2111048. PMID 12153968
- [Background] Rappaport EB, Gilliland FD, Linn WS, Gauderman WJ. Impact of respiratory illness on expiratory flow rates in normal, asthmatic, and allergic children. Pediatr Pulmonol. 2002 Aug;34(2):112-21. doi: 10.1002/ppul.10142. PMID 12112777
- [Background] Gilliland FD, Berhane KT, Li YF, Kim DH, Margolis HG. Dietary magnesium, potassium, sodium, and children's lung function. Am J Epidemiol. 2002 Jan 15;155(2):125-31. doi: 10.1093/aje/155.2.125. PMID 11790675
- [Background] Gilliland FD, Li YF, Peters JM. Effects of maternal smoking during pregnancy and environmental tobacco smoke on asthma and wheezing in children. Am J Respir Crit Care Med. 2001 Feb;163(2):429-36. doi: 10.1164/ajrccm.163.2.2006009. PMID 11179118
- [Background] Gilliland FD, Berhane K, Rappaport EB, Thomas DC, Avol E, Gauderman WJ, London SJ, Margolis HG, McConnell R, Islam KT, Peters JM. The effects of ambient air pollution on school absenteeism due to respiratory illnesses. Epidemiology. 2001 Jan;12(1):43-54. doi: 10.1097/00001648-200101000-00009. PMID 11138819
- [Background] Li YF, Gilliland FD, Berhane K, McConnell R, Gauderman WJ, Rappaport EB, Peters JM. Effects of in utero and environmental tobacco smoke exposure on lung function in boys and girls with and without asthma. Am J Respir Crit Care Med. 2000 Dec;162(6):2097-104. doi: 10.1164/ajrccm.162.6.2004178. PMID 11112121
- [Background] Gilliland FD, Berhane K, McConnell R, Gauderman WJ, Vora H, Rappaport EB, Avol E, Peters JM. Maternal smoking during pregnancy, environmental tobacco smoke exposure and childhood lung function. Thorax. 2000 Apr;55(4):271-6. doi: 10.1136/thorax.55.4.271. PMID 10722765
- [Background] Gilliland F, Avol E, Kinney P, Jerrett M, Dvonch T, Lurmann F, Buckley T, Breysse P, Keeler G, de Villiers T, McConnell R. Air pollution exposure assessment for epidemiologic studies of pregnant women and children: lessons learned from the Centers for Children's Environmental Health and Disease Prevention Research. Environ Health Perspect. 2005 Oct;113(10):1447-54. doi: 10.1289/ehp.7673. PMID 16203261